CLINICAL TRIAL: NCT05860335
Title: Efficacy and Safety ofToripalimab Combined With AP-induced Chemotherapyfollowed by Concurrent Chemoradiotherapy and Toripalimab-maintenance Therapysequentially in Patients With Non-metastatic IVB Hypopharyngeal Cancer : Aopen-lablc, Single-arm ,Phase II Clinical Study
Brief Title: Efficacy and Safety of Toripalimab Combined With AP-induced Chemotherapy Followed in Non-metastatic IVB Hypopharyngeal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Xinxin Zhang, Director, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Interventional
Record Dates: First submitted 2023-04-24; First posted 2023-05-16 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Hypopharyngeal Cancer
Keywords: non-metastatic IVB hypopharyngeal cancer; Toripalimab; Combine therapy
MeSH Terms: conditions — Hypopharyngeal Neoplasms | interventions — Cisplatin; nedaplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Toripalimab +AP-induced chemotherapy (Experimental): Study drug: toripalimab JS001 dosage：240mg Drug administration plan and mode：Intravenous infusion of 30min (not less than 20min and not more than 60min), followed by observation of 60min (only the first 2 cycles), once every 3 weeks (Q3W).
  Interventions: Drug: Cisplatin/Nedaplatin, albumin paclitaxel

INTERVENTIONS:
Drug: Cisplatin/Nedaplatin, albumin paclitaxel — During induction chemotherapy, triplelimab JS001 was administered before cisplatin/Nedaplatin and albumin paclitaxel. JS001 Intravenous infusion of cisplatin/Nedaplatin was administered 60 minutes after the end of infusion and beginning on day 1 of each cycle 40mg/m 2, D1, D2 albumin paclitaxel 230 mg/m 2; Chemotherapeutic drugs are administered in accordance with the drug label and local prodrome and other standard protocols for prophylactic use, every 3 Once a week (Q3W) for 2 cycles

SUMMARY:
The goal of this type of study: single center exploratory clinical trial is to evaluate the efficacy and safety of Toripalimab combined with AP-induced chemotherapy followed by concurrent chemoradiotherapy and Toripalimab-maintenance therapy sequentially in patients with non-metastatic IVB hypopharyngeal cancer. The main question[s] it aims to answer are: • [main objectives: to evaluate the objective remission rate (ORR), progression-free survival (PFS) and safety of PD-1 inhibitor Toripalimab combined with induction chemotherapy (cisplatin / nedaplatin + albumin paclitaxel) in patients with locally advanced head and neck squamous cell carcinoma according to RECISTv1.1.] • [Secondary objectives: 1-year, 2-year, 3-year progression-free survival rate (PFS); 1-year, 2-year, 3-year overall survival rate (OS); overall survival time (OS); tumor regression time; quality of life was evaluated by ECOG physical status and EQ-5D-5L assessment. ] [Exploratory Objective: to explore the relationship between the biomarkers in tumor tissue and / or blood, including PD-L1 (CPS/TPS), HPV (P16), PD-1, TMB, EGFR, CD3, CD4, CD8, TP53, MSI-H and the efficacy of immunotherapy, and the relationship between MDM2/MDM4, EGFR, chromosome 11q13 interval (CCND1/FGF19/FGF3/FGF4) and immune hyperprogression] Participants will [be treated with Toripalimab injection (240mg/, once every 3 weeks) combined with cisplatin / nedaplatin (40mg) and albumin paclitaxel (230mg/m2, once every 3 weeks). The efficacy was evaluated within 1 week after induction therapy. In the phase of simultaneous radiotherapy, albumin paclitaxel (230mg/m2, once every 3 weeks, D1/D21/D43) was used. One month after the end of synchronous radiotherapy and chemotherapy, the efficacy was evaluated. After evaluation, all patients entered the next stage of immune maintenance therapy. During the maintenance phase, Toripalimabv injection (240mg/, once every 3 weeks) was given for 6 months or until the disease progressed, the toxicity was intolerable, the subjects asked to withdraw voluntarily, and the researchers judged that the subjects needed to withdraw from the study. The patients were treated with spiral tomographic radiotherapy (TOMO) or intensity modulated radiotherapy (IMRT).. These patients were given Nimotuzumab injection at the same time during simultaneous radiotherapy and chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 70 years old
2. The clinical stage was Ivb stage (AJCC 8th edition),
3. ECOG score was 0-1
4. Have not received any anti-tumor therapy such as radiotherapy, chemotherapy, immunotherapy or biological therapy
5. No contraindications of chemotherapy, immunotherapy and radiotherapy
6. The functional level of major organs conforms to the following criteria: 1) the standard of blood routine examination should meet the following criteria: WBC ≥ 3.0x109, G-CSF and other hematopoietic stimulating factors. 2) biochemical tests should meet the following criteria: TBIL ≤ 2.0 × ULN,ALT, AST ≤ 2.5 × ULN,BUN and CRE ≤ 1.5 × ULN or endogenous creatinine clearance ≥ 60ml/min (Cockcroft-Gault formula); 3) good coagulation function: defined as international standardized ratio (INR) or prothrombin time (PT) ≤ 1.5 times ULN; if the subject is receiving anticoagulant therapy, as long as PT is within the range of anticoagulant use. 4) Myocardial zymogram is within the range of normal value;
7. Women of childbearing age must have taken reliable contraceptive measures, or conducted pregnancy tests (serum or urine) within 7 days before admission, and the results were negative, and were willing to use effective methods of contraception during the trial period and within 2 months after the last administration of anti-PD-1 antibody. For male subjects whose partners are women of childbearing age, effective methods of contraception should be used during the trial and within 2 months after the last administration of anti-PD-1 antibody. 8. The subjects voluntarily joined the study, signed the informed consent form, had good compliance and cooperated with follow-up.

Exclusion Criteria:

1. Previous or simultaneous suffering from other uncured malignant tumors, except cured basal cell carcinoma of the skin, carcinoma in situ of the cervix and superficial bladder cancer
2. Patients with hypopharyngeal necrosis at the same time with the risk of bleeding.
3. Suffer from any active autoimmune disease or have a history of autoimmune disease (e.g. interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism (can be included when hormone replacement therapy is normal). Patients with vitiligo or asthma who have been completely relieved in childhood and can be included after adulthood without any intervention, and asthma patients who need bronchodilators for medical intervention can not be included.
4. Suffering from uncontrolled cardiovascular disease: myocardial ischemia or myocardial infarction of grade Ⅱ or above, poorly controlled arrhythmias (including QTc interval ≥ 470ms); cardiac insufficiency of grade Ⅲ ~ IV according to NYHA criteria, or left ventricular ejection fraction (LVEF) < 50% indicated by color Doppler ultrasound; myocardial infarction occurred within 1 year.
5. There is an active infection or an unexplained fever occurs during the screening period and before the first administration of the drug > 38.5 ℃ (according to the researchers, the fever caused by the tumor can be included in the group).
6. Suffer from congenital or acquired immune deficiency (such as HIV infection), active hepatitis B (HBV-DNA ≥ 104copies / ml) or hepatitis C (hepatitis C antibody positive and HCR-RNA higher than the lower limit of detection by analytical method).
7. Have previously received other PD-1 antibody therapy or other immunotherapy for PD-1/PD-L1.
8. Known to be allergic to paclitaxel, cisplatin, macromolecular protein preparations, or any anti-PD-1 antibody component.
9. If the subject has undergone a major operation, the toxic reactions and / or complications caused by the surgical intervention must be fully recovered before starting the treatment.
10. Within 4 weeks before the first use of research drugs (subjects who have entered the follow-up period are calculated on the basis of their last use of experimental drugs or devices) or are participating in other clinical studies.
11. Live vaccine and COVID-19 vaccine are given within 4 weeks before the first use of the study; inactivated virus vaccine for seasonal influenza is allowed; live attenuated influenza vaccine for nasal use is not allowed.
12. Pregnant or lactating women.
13. The researchers determined that the subjects had other factors that might force them to stop the study, such as other serious illnesses (including mental illness) requiring combined treatment, seriously abnormal laboratory tests, family or social factors, which may affect the safety of the subjects or the collection of trial data.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate （ORR） | 3 years
  An objective response is defined as either a confirmed CR or a PR, as determined by the investigator using RECIST v1.1Response Evaluation Criteria in Solid Tumors (RECIST) from the National Cancer Institute (NCI).
Progress-free survival (PFS) | 1years， 2 years ， 3 years
  Defined from date of randomization to date of first documentation of progression or death due to any cause For example, increased tumor burden (including new small lesions in non critical areas), physical fitness status, and experimentation If there is no significant deterioration in the room value, treatment is allowed to continue until at least 4 weeks later or the next planned period Repetitive imaging examination confirms disease progression at the time point of imaging examination
Incidence rate of adverse events (AEs) | 3 years
  Analysis of adverse events (AEs) are based on treatment-related AEs (trAEs) and immune-related AEs (irAEs), and all-grade AEs and grade 3-4 AEs. AEs are evaluated by investigators according to the Common Terminology Criteria for Adverse Events, version 5.0

SECONDARY OUTCOMES:
Overall survival (OS) | 1years， 2 years ， 3 years
  Defined from date of randomization to date of first documentation of death from any cause or censored at the date of the last follow-up.
ECOG physical fitness status | Once a week for the duration of treatment, 15, 18, 21, and 24 months after completion of treatment
  The physical condition of patients in the evaluation group was evaluated by ECOG score
Tumor regression time | 3 years
Quality of Life (QOL) | 3 years
  Evaluate the quality of life of patients in the evaluation group through EQ-5D-5L assessment

CONTACTS AND LOCATIONS:
Locations (1):
- 中国人民解放军总医院, Beijing, China